CLINICAL TRIAL: NCT06280235
Title: A Phase II, 6-week, Multicenter, Randomized, Double Blind (Patient and Investigator) or Masked, Placebo Controlled, Dose-finding Trial to Evaluate the Efficacy, Tolerability, and Safety of Different Doses of Oral BI 1569912 as Adjunctive Therapy in MD
Brief Title: A Study to Test Different Doses of BI 1569912 in People With Depression Who Take Anti-depressive Medicine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1447-0005; U1111-1297-3126 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2023-507942-10-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 1569912 low dose group (Experimental)
  Interventions: Drug: BI 1569912
- BI 1569912 medium dose group (Experimental)
  Interventions: Drug: BI 1569912
- BI 1569912 high dose group (Experimental)
  Interventions: Drug: BI 1569912
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: BI 1569912 high dose group; BI 1569912 low dose group; BI 1569912 medium dose group
Drug: Placebo — Placebo matching BI 1569912
  Arms: Placebo group

SUMMARY:
This study is open to adults between 18 and 65 with a type of depression (major depressive disorder) for whom previous treatments for depression did not work. The purpose of the study is to find out whether a medicine called BI 1569912 helps people with depression.

Participants continue their standard therapy throughout the study.

Participants are put into 4 groups by chance. 3 of the 4 groups take different doses of BI 1569912. 1 group takes placebo. Placebo tablets looks like BI 1569912 but do not contain any medicine. Participants take the tablets once a day for 6 weeks.

Participants are in the study for about 2 to 4 and a half months. During this time, they visit the study site at least 6 times. At the visits, doctors ask participants about their symptoms.

The participants answer questions about their depression symptoms. The results are compared between the groups. The doctors also regularly check the general health of participants.

ELIGIBILITY:
Inclusion criteria:

1. Male and female participants, 18 to 65 years of age, both inclusively at the time of consent.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Women of childbearing potential (WOCBP) must be ready and able to use a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly plus one additional barrier method. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information and in the study protocol.
4. Established diagnosis of major depressive disorder (MDD), single episode or recurrent, as confirmed at the time of screening by the mini-international neuropsychiatric interview (MINI) with a duration of current depressive episode ≥8 weeks at the time of screening visit.
5. Hamilton Depression Rating Scale-17 (HDRS-17) - Severity scale score >17.
6. A documented ongoing monotherapy treatment of ≥6 weeks at the randomisation visit, with an selective serotonin reuptake inhibitor (SSRI) or serotonin and norepinephrine reuptake inhibitor (SNRI) specified in the investigator site file (ISF) at adequate dose (at least minimum effective dose as per prescribing information).

   * The participant must adhere to the screening visit dose of the background SSRI/SNRI until the end of the trial. Participants should be on a stable dose for at least 4 weeks prior to randomisation.
   * Participants, who, in addition to their monotherapy with an SSRI/SNRI, are taking additional low dose antidepressant medications for purposes other than treating depressive symptoms, are not excluded. The dose must be less than the lowest dose indicated for MDD.
7. In the current episode, participants have shown insufficient treatment response defined by less than 50% response to a maximum of 4 antidepressant treatments of adequate dose and treatment duration (according to Summary of Product Characteristics) as evaluated by the antidepressant treatment response questionnaire (ATRQ).

Exclusion criteria:

1. Per MINI, have ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, or delusional disorder.
2. Diagnosis with antisocial, paranoid, schizoid or schizotypal personality disorder, or MDD with psychotic features as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria, at the time of screening visit. Any other personality disorder at screening visit that significantly affects current psychiatric status and likely to impact trial participation, as per the judgement of investigator.
3. Diagnosis of any other mental disorder that was the primary focus of treatment within 6 months prior to screening (as per clinical discretion of the investigator).
4. History or presence (upon clinical examination) of seizure disorders or an increased risk of seizures (first degree relative with epilepsy), stroke, brain tumour or any other major neurological illness that could impact participation in the trial.
5. A current or recent history of clinically significant suicidal ideation with intent within the past 3 months, corresponding to a score of 4 or 5 for ideation on the Columbia-suicide severity rating scale (C-SSRS) or a suicidal attempt within the past year, as indicated by the C-SSRS at screening visit.
6. Participants with a body mass index (weight [kg]/height [m]²) lower than 18 kg/m² or greater than 40 kg/m² at screening.
7. Diagnosis of a moderate to severe substance related disorder within 6 months prior to screening visit (with exception of caffeine and tobacco).
8. Positive drug screen (amphetamines, opiates, cocaine, barbiturates, phencyclidine) at screening or Visit 1A (if applicable). Participants with positive cannabis and benzodiazepine drug tests can be included if the investigator confirms that there is no active substance related disorder. Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) total score at Week 6 | at baseline, at week 6
  The MADRS evaluates core symptoms of depression. It is a clinician-rated measure of depression severity and consists of 10 items. MADRS items are rated on a 0-6 continuum (0 = no abnormality, 6 = severe).
  The possible total score could range from 0 to 60 - from normal with absence of symptoms to severe depression.

SECONDARY OUTCOMES:
Change from baseline in MADRS total score at Day 8 | at baseline, at day 8
Response defined as ≥50% MADRS reduction from baseline at Day 8 | at baseline, at day 8
Response defined as ≥50% MADRS reduction from baseline at Week 6 | at baseline, at week 6
Remission defined as MADRS total score ≤10 at Week 6 | up to 6 weeks
Change from baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) total score at Day 8 | at baseline, at day 8
  The SMDDS is a 16-item, patient-reported outcome (PRO) measure developed to capture the core symptoms of major depressive disorder (MDD).
  Participants respond to each question using a rating scale between 0 ("Not at all" or "Never") to 4 ("Extremely" or "Always").
  The total score ranges from 0 to 60 with a higher score indicating more severe depressive symptomatology.
  It is calculated by creating first a single score for items 11 and 12 by selecting the highest severity on either item, and then creating the sum of the 15 responses.
Change from baseline in SMDDS total score at Week 4 | at baseline, at week 4

CONTACTS AND LOCATIONS:
Locations (53):
- United States (22):
  - Southwest Biomedical Research, LLC, Tucson, Arizona
  - Excell Research Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers-Panorama City-62905, Panorama City, California
  - CT Clinical Research, Cromwell, Connecticut
  - Galiz Research, Hialeah, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - CCM Clinical Research Group, LLC-Miami-68482, Miami, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Chicago Research Center, Incorporated, Chicago, Illinois
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Boston Clinical Trials, Roslindale, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Hassman Research Institute-Marlton-66897, Marlton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Midwest Clinical Research, Dayton, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Belgium (2):
  - Anima Research Center, Alken
  - Universitair Psychiatrisch Centrum Duffel (UPC Duffel), Duffel
- Bulgaria (7):
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry - Dr Ivo Natsov, Cherven Bryag
  - MHC - Ruse, EOOD, Rousse
  - Medical Center "Sv.Naum", Sofia
  - DCC "Sv. Vrach and Sv. Sv. Kuzma and Damyan" OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica Ltd., Sofia
  - DCC Mladost-M Varna OOD, Varna
- China (8):
  - Hebei Mental Health Center, Baoding
  - Beijing Anding Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - Shanghai Mental Health Center, Shanghai
  - Shenzhen Kangning Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
- Czechia (2):
  - A-SHINE s.r.o, Pilsen
  - Clintrial s.r.o., Prague
- Germany (2):
  - Charite Universitätsmedizin Berlin KöR, Berlin
  - Somni Bene - Institut für Medizinische Forschung & Schlafmedizin Schwerin GmbH, Schwerin
- Japan (10):
  - Iwaki Clinic, Tokushima, Psychosomatic Medicine, Anan-shi
  - Aisakura Clinic, Fukuoka
  - Kaku Mental Clinic, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Rainbow and Sea Hospital, Karatsu-shi
  - Hirota Clinic, Kurume-shi
  - Kyorin University Hospital, Mitaka-shi
  - Maynds Tower Mental Clinic, Shibuya-ku

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com